CLINICAL TRIAL: NCT03935061
Title: Auxiliary Effects of Mulberry Juice on Inflammatory Status and Clinical Symptoms in Patients With General Anxiety Disorder: A Single-Blinded Trial
Brief Title: Effects of Mulberry Juice on Inflammatory Status and Clinical Symptoms in Patients With General Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201802079
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-04

CONDITIONS: General Anxiety Disorders; Systemic Inflammation; Interleukin
Keywords: Anthocyanin; Anxiety Disorders; Inflammation; interleukin-17A
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders; Inflammation

STUDY DESIGN:
Intervention Model Description: Patients who agree to join our study are measured at baseline. Randomization is carried out by using a computer program and 2 bottles (600 ml/bottle) of sanitized mulberry juice are delivered to the experimental group 20 days before the next clinic visit, with instruction to consume 50 ml of juice diluted with drinking water at room temperature. For the control group, patients are informed of their allocation results along with a reminder of the next clinic visit. On the second visit at the 1st month, measurements of clinical symptoms and social functions and inflammation status are conducted. A between-group difference at this stage represents changes caused by the intervention. No mulberry juice is given to patients for either group further on. All patients are evaluated again with the same assessment tools, as well as the immunology markers in their sera during the third visit.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinical assessments of clinical symptoms and social functions are self-reported and thus clinicians or care providers have no knowledge of the outcomes. The self-reported assessments are then coded by a research assistant with masked group labels and handled to the statistician for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulberry juice (Experimental): Two bottles (600 ml/bottle) of sanitized mulberry juice are delivered to the patients of the experimental group 20 days before the next clinic visit, with instruction to consume 50 ml of juice diluted with drinking water at room temperature. A reminder of the next clinic visit for continuous treatment is attached.
  Interventions: Other: Mulberry juice
- Controlled (No Intervention): Patients of the controlled group are informed of their allocation results along with a reminder of the next clinic visit. On the second visit at the 1st month, measurements of clinical symptoms and inflammation status are conducted. No mulberry juice is given to patients further on. All patients are evaluated again with the same assessment tools, as well as the immunology markers in their sera during the third visit.

INTERVENTIONS:
Other: Mulberry juice — On the second visit at the 1st month, measurements of clinical symptoms and inflammation status are conducted. No mulberry juice is given to patients further on. All patients are evaluated again with the same assessment tools, as well as the immunology markers in their sera during the third visit.
  Arms: Mulberry juice

SUMMARY:
Anxiety and depression are normally associated with inflammation reactions and interleukin (IL) related pathways are most evidently involved. IL-17A (interleukin 17A) induces psoriasis-like inflammation and depression-like behaviors in animals and can be relieved by using IL-17A antibody. Also, human association studies found that IL-17A and certain downstream ILs are associated with the severity of anxiety. IL-17A is a sentinel cytokine. On binding with interleukin 17A receptor (IL-17RA) and interleukin 17C receptor (IL-27RC), it induces signaling cascades via nuclear factor kappa-light-chain-enhancer of activated B cells (NFκB), P38 mitogen-activated protein kinases (p38MAPK) and CCAAT-enhancer-binding proteins (C/EBPs) knots, and stimulates subsequent cell secretions of cytokines and chemokines. Cyanidin 3-O-glucoside, the main anthocyanin component of mulberry, competes with IL-17A to bind its receptors and inhibits subsequent downstream cascades. The investigators plan to use a single-blinded randomized controlled trial to evaluate the auxiliary effect of mulberry juice in general anxiety disorder, including differences in psychiatric symptoms and levels of IL-related markers between the experimental and control groups, and contribution of IL-related genes in the auxiliary effect.

DETAILED DESCRIPTION:
The etiology, pathogenesis, and pathophysiology of psychiatric disorders are not limited to the brain. Anxiety and depression are normally associated with inflammation reactions and interleukin (IL) related pathways are most evidently involved. Previous animal studies showed that administration of IL-17A induces psoriasis-like inflammation and depression-like behavior, and can be relieved by using IL-17A antibody, while in humans, association studies showed that serum IL-17A and certain downstream ILs are associated with the severity of anxiety. Also, the result of human genetic studies also identified several IL genes associated with anxiety and depression. IL-17A is a sentinel cytokine. On binding with interleukin 17A receptor (IL-17RA) and interleukin 17C receptor (IL-27RC), it induces signaling cascades via nuclear factor kappa-light-chain-enhancer of activated B cells (NFκB), P38 mitogen-activated protein kinases (p38MAPK) and CCAAT-enhancer-binding proteins (C/EBPs) knots, and stimulates subsequent cell secretions of cytokines and chemokines. Many studies have demonstrated that consumption of proanthocyanidin-rich or anthocyanin-rich berries, berries juice or other secondary products reduce a variety of inflammation symptoms in humans. However, these berries do not meet a low-cost requirement for general nutritional recommendation and new drug development in Taiwan due to the additional import cost. On the other hand, cyanidin 3-O-glucoside, the main anthocyanin component of local mulberry, competes with IL-17A to bind its receptors and inhibits subsequent downstream cascades. Without interfering the on-going treatment of the patients, this proposal plans to use a single-blinded randomized controlled trial to evaluate the auxiliary effect of mulberry juice in general anxiety disorder, including differences in psychiatric symptoms (anxiety, depression, and functions) and levels of IL-related markers between the experimental and control groups, and contribution of IL-related genes in the auxiliary effect.

ELIGIBILITY:
Inclusion Criteria:

• meet the criteria for GAD in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, as their primary diagnosis

Exclusion Criteria:

* severe physical diseases that required intensive care or additional medical attention such as terminal cancer, stroke, and end-stage renal disease
* psychotic symptoms or recent suicide attempts

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
General Anxiety Disorder-7 items (GAD-7) | 5 to 10 minutes
  GAD-7 measures anxiety status. The questionnaire is self-reported.
Patient Health Questionnaire-9 items (PHQ-9) | 5 to 10 minutes
  PHQ-9 measure depression status. This questionnaire is self-reported.
World Health Organization Quality of Life - Brief (WHOQOL-BREF) | 5 to 10 minutes
  WHOQOL-BREF measures the quality of life. The questionnaire is self-reported.

SECONDARY OUTCOMES:
Inflammation markers | 6 months
  Inflammation status of the patients are evaluated by measuring CRP, known cytokines (Interleukin- 6 [IL-6], Interleukin-1β [IL-1β], tumor necrosis factor-α (TNF-α), granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF], and transforming growth factor [TGF-β]), chemokines (IL-8, GRO-α, and MCP-1), and PGE in sera, in addition to the sentinel molecule IL-17A. All markers are measured by using ELISA assays according to manufacturer instructions.
Inflammation genes | 24 months
  Inflammation genes including CRP, cytokines (IL-6, IL-1β, TNF-α, G-CSF, GM-CSF, and TGF-β), chemokines (IL-8, GRO-α, and MCP-1), and PGE in addition to IL-17A, are to be genotyped.

CONTACTS AND LOCATIONS:
Overall Officials: El-Wui Loh, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan